CLINICAL TRIAL: NCT00561210
Title: Effect of Early Enteral Tube Feeding Nutrition With an Immune Enhancing Diet in Severe Burn Patients
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Société des Produits Nestlé (SPN) (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: NCNF 0501
Record Dates: First submitted 2007-11-16; First posted 2007-11-20 (Estimated); Last update posted 2013-11-19 (Estimated); Status verified 2013-11

CONDITIONS: Infections on; Severe Burn Patients
Keywords: infections
MeSH Terms: conditions — Infections

ARMS (2):
- I (Experimental): Total enteral tube feeding
  Interventions: Dietary Supplement: Crucial
- II (Active Comparator): Total enteral tube feeding
  Interventions: Dietary Supplement: Sondalis HP

INTERVENTIONS:
Dietary Supplement: Crucial — Treatment between minimum 14 days and maximum 6 months. Apports depend on method of CURRERI.
  Arms: I
Dietary Supplement: Sondalis HP — Treatment between minimum 14 days and maximum 6 months. Apports depend on method of CURRERI.
  Arms: II

SUMMARY:
Compare clinical and biological effects of two enteral tube feeding nutrition formula (immune enhancing diet versus polymeric diet)in severe burn hospitalized patients .

ELIGIBILITY:
Inclusion Criteria:

* Thermic burn from 20% to 80%
* 15 < age < 70 years
* written informed consent

Exclusion Criteria:

* diabetes mellitus
* corticoid or immuno-suppressive therapy
* HIV
* evolutive cancers
* pregnancy
* abdominal lesion
* hepatic or renal failure

Ages: 15 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 57 (Actual)
Dates: Start 2003-11; Primary Completion 2010-03 (Actual); Study Completion 2010-03 (Actual)

PRIMARY OUTCOMES:
Number of infections and number of multiple organ failure | 6 months

SECONDARY OUTCOMES:
digestive tolerance and healing | 6 months

CONTACTS AND LOCATIONS:
Overall Officials: Cecile Chambrier, Study Chair — Hopital Edouard Herriot - Lyon
Locations (5):
- France (5):
  - CHU Pellegrin-Unites des brules, Bordeaux
  - Hôpital Saint Luc - Service des brûlés, Lyon
  - Hôpital Edouard Herriot, Lyon
  - Hopital Hotel Dieu-Service des brules, Nantes
  - Hopital Saint Antoine- Service des Brules, Paris